CLINICAL TRIAL: NCT05864781
Title: The Effect of Jigsaw Technique Used in Critical Article Review Given by Distance Education on Critical Thinking Disposition and Communication Skills of Nursing Students - Quasi-Experimental Study
Brief Title: The Effect of Jigsaw Technique Used in Critical Article Review on Critical Thinking Disposition and Communication Skills
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duzce University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: DuzceU-merve-0001
Record Dates: First submitted 2023-05-09; First posted 2023-05-18 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Education, Distance; Students, Nursing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): With the students in the control group, a standard individual article review will be conducted under the supervision of the instructor.
- Experimental group (Experimental): The students in the experimental group will be divided into 8 main groups of 7 students according to their academic grade point average. In these groups, each member will be responsible for one of the 7 sections of the article. Those who take the same section in the groups will unite to form expert groups and specialize by working on this section. Students will then return to their main groups and analyze an experimental article. From the groups presenting their reviews, a winner will be selected and a prize will be awarded.
  Interventions: Behavioral: Jigsaw Technique

INTERVENTIONS:
Behavioral: Jigsaw Technique — Jigsaw technique is one of the cooperative learning methods. A topic planned to be learned in the lesson is divided into sections and these sections are distributed to the students in the main group. Students who are responsible for the same sections in the groups combine to form expert groups and specialize by working on the subject. They then return to their main group to share their knowledge and make a presentation on the topic.
  Arms: Experimental group

SUMMARY:
For nursing education to be sufficient to provide students with the contemporary roles required by the profession, education programs should be provided that will enable students to participate in the learning-teaching process actively. One of these programs is cooperative learning methods. The jigsaw learning technique, one of the collaborative learning methods, creates a contemporary learning model by providing a positive learning environment, individualization of students and the development of a sense of responsibility. Since distance education has become widespread worldwide, it is necessary to use these methods to increase interaction and group work in distance education.

Aim: This study aims to determine the effect of the Jigsaw technique used in critical article reviews given by distance education on the critical thinking disposition and communication skills of nursing students.

DETAILED DESCRIPTION:
For nursing education to be sufficient to provide students with the contemporary roles required by the profession, education programs should be provided that will enable students to participate in the learning-teaching process actively. One of these programs is cooperative learning methods. The jigsaw learning technique, one of the collaborative learning methods, creates a contemporary learning model by providing a positive learning environment, individualization of students and the development of a sense of responsibility. Since distance education has become widespread worldwide, it is necessary to use these methods to increase interaction and group work in distance education.

Aim: This study aims to determine the effect of the Jigsaw technique used in critical article reviews given by distance education on the critical thinking disposition and communication skills of nursing students.

Method: This is a quasi-experimental study. The study will be carried out in the Spring Semester of the 2022-2023 Academic Year, with the students who attend the Research in Nursing Course with distance education at the Nursing Department of the Faculty of Health Sciences of Duzce University. The study is planned to comprise 112 students, 56 students in each group, taking into account possible losses. The sample was calculated using the G*Power 3.1.9.7 programme.

Data accumulation methods: In the study, descriptive features form, critical thinking disposition scale and communication skills scale will be used as data collection tools.

Pre-tests will be administered to the students in the control group after the theoretical part of the course is over. Individual homework will be given to the students and they will be provided to analyze articles under the supervision of the researcher. Post-tests will be applied.

Students in the experimental group will be administered a pre-test. Students will be heterogeneously divided into eight groups according to their academic grade point average. The groups will consist of 7 people. Each student will be responsible for one of the 7 article sections. These sections are: 1) Title - Abstract 2) Introduction 3) Method 4) Results 5) Discussion 6) Conclusion and Recommendations 7) Limitations - Resources. Within the group, it will be determined which member will be responsible for which article section.

Students who have chosen the same article section in their main groups will come together to form expert groups. These expert groups are called "Peer critical article review" groups. After the expert groups are determined, they will come together and learn the article section they will be experts on. To ensure positive group cohesion during the group process in expert group work, members will be assigned one of the responsibilities of group leader, reporter, and monitoring the participation of members. The researcher will answer the questions asked by the students during the expert group work and provide support to the groups (3 hours).

Students who are experts in their chosen article section return to their main groups to share their knowledge. Each group reviews one descriptive research and presents their review (3 hours). The instructor advises and selects the first group. The first group wins a research award with the support of the lecturers.

Experiences in the process are shared and Post-tests are applied.

ELIGIBILITY:
Inclusion Criteria:

* Students must volunteer to participate in the study.

Exclusion Criteria:

* Students who decline to participate in the study
* Students who will not be able to participate in the application continuously

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 112 (Estimated)
Dates: Start 2023-05-12 (Actual); Primary Completion 2025-06-12 (Estimated); Study Completion 2025-08-12 (Estimated)

PRIMARY OUTCOMES:
Critical Thinking Disposition | 28 to 30 days
  Critical Thinking Disposition Scale: The scale was developed by Semerci in 2000. The scale consists of 49 items with 5 dimensions. Sub-themes of the scale are metacognition, flexibility, systematicity, tenacity-patience and open-mindedness. 14 of the items are in metacognition, 11 of these are in flexibility, 11 of these are in tenacity-patience, and 8 of these are in open-mindedness. Scale defines how students perceive interpretation, analysis, inference, and evaluation from a reasoned point of view. The evaluation of the scale is performed over each sub-scale and the total score of the scale. Cronbach Alpha coefficient of the Critical Thinking Disposition is 0.96.
Communication Skills | 28 to 30 days
  The Communication Skills Scale helps to determine the communication skills of the students. Scale items centred on the factors of "competence", "discouragement", "body language" and "dignification" factors and there were 36 items in total. The lowest score that can be obtained from the entire scale is 36 and the highest score is 180. In the sub-dimensions of the scale, the lowest score that can be obtained from the competence dimension is 12, the highest score is 60; The lowest score that can be obtained from the disability dimension is 13, and the highest score is 65; The lowest score that can be obtained from the body language dimension is 5, the highest score is 25; The lowest score that can be obtained from the valuing dimension is 6 and the highest score is 30 points. It can be concluded that as the scores obtained from the scale increase, the level of communication skills also increases. Cronbach's alpha coefficient of the scale is 0.89.

CONTACTS AND LOCATIONS:
Overall Officials: Merve Cakar, PhD, Principal Investigator — Duzce University
Locations (1):
- Duzce University, Düzce, Turkey (Türkiye)